CLINICAL TRIAL: NCT04439851
Title: The Relationship Between Monocyte-to-High-Density Lipoprotein Cholesterol Ratio, Metabolic Parameters and Excess Weight Loss in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Impact of Sleeve Gastrectomy on Monocyte-to-High-Density Lipoprotein Cholesterol Ratio
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sibel Ocak Serin, Principal Investigator, Umraniye Education and Research Hospital
Other Study IDs: umraniye training hospital
Record Dates: First submitted 2020-06-10; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Laparoscopic Sleeve Gastrectomy; Cardiovascular Risk Factor; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study hypothesized that significant weight loss is associated with a reduction in the inflammatory markers, leading to diminished cardiovascular risks in patients undergoing laparoscopic sleeve gastrectomy (LGS).

We found a decrease in MHR at postoperative 6 months from baseline in patients undergoing LSG. The decrease in MHR was more remarkable with increasing percentage of EWL, but no relationship between the %EWL and MHR.

DETAILED DESCRIPTION:
The present study aims to evaluate the relationship between MHR, metabolic parameters and the percentage of excess weight loss (%EWL) in participants undergoing laparoscopic sleeve gastrectomy (LSG).

This prospective cohort study will evaluate obese participants undergoing LSG. Demographic data of the participants and blood glucose level, monocyte count and lipid parameters baseline and at 6 months after surgery will record. The MHR baseline and at 6 months after surgery and the %EWL at 6 months after surgery will calculate. The participants will be divide into two groups as participants with %EWL of <50 and patients with a %EWL of ≥50. The parameters will compare between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Obese patients (BMI ≥40 or >35+ and accompanying DM, HT and hyperlipidemia) Underwent laparoscopic sleeve gastrectomy.

Exclusion Criteria:

Receiving antihyperlipidemic therapy, Important complications that continue within 6 months after surgery (anastomotic leaks, pulmonary embolism, deep vein thrombosis, soft tissue infection) Did not attend 6-month control visit were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients (BMI ≥40 or >35+ and accompanying DM, HT and hyperlipidemia)
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Monocyte-to-High-Density Lipoprotein Cholesterol Ratio changes | 6 months
  Monocyte-to-High-Density Lipoprotein Cholesterol Ratio changes after Sleeve Gastrectomy